CLINICAL TRIAL: NCT03490162
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Pharmacokinetics of Single and Multiple Ascending Doses and Effect of Food on the Pharmacokinetics of DM1157 in Healthy Adults
Brief Title: Safety and Pharmacokinetics Study of DM1157 to Treat Malaria
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: There was toxicity in higher dose groups and a therapeutic dose level was not found in lower dose groups.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0088; HHSN272201500006I
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2019-04-30

CONDITIONS: Malaria
Keywords: Anti-Malarial; DM1157; Pharmacokinetics; Safety
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Food Effect (Experimental): 300 mg of DM1157 (2 capsules of 150 mg) orally with high fat diet, n=6, and matching placebo (2 capsules) orally with high fat diet, n=2
  Interventions: Drug: DM1157; Other: Placebo
- MAD 1 (Experimental): 150 mg of DM1157 (1 capsule) orally daily for three days with 240 ml of water after an overnight fast, n=8, and matching placebo (1 capsule) orally daily for three days with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- MAD 2 (Experimental): 300 mg of DM1157 (2 capsules of 150 mg) orally daily for three days with 240 ml of water after an overnight fast, n=8, and matching placebo (2 capsules) orally daily for three days with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- MAD 3 (Experimental): 600 mg of DM1157 (4 capsules of 150 mg) orally daily for three days with 240 ml of water after an overnight fast, n=8, and matching placebo (4 capsules) orally daily for three days with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- MAD 4 (Experimental): 900 mg of DM1157 (6 capsules of 150 mg) orally daily for three days with 240 ml of water after an overnight fast, n=8, and matching placebo (6 capsules) orally daily for three days with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- SAD 1 (Experimental): 9 mg of DM1157 (1 capsule) orally with 240 ml of water after an overnight fast, n=6, and matching placebo (1 capsule) orally with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- SAD 2 (Experimental): 27 mg of DM1157 (3 capsules of 9 mg) orally with 240 ml of water after an overnight fast, n=6, and matching placebo (3 capsules) orally with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- SAD 3 (Experimental): 81 mg of DM1157 (9 capsules of 9 mg) orally with 240 ml of water after an overnight fast, n=6, and matching placebo (9 capsule) orally with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- SAD 4 (Experimental): 150 mg of DM1157 (1capsule) orally with 240 ml of water after an overnight fast, n=6, and matching placebo (1 capsule) orally with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- SAD 5 (Experimental): 300 mg of DM1157 (2 capsules of 150 mg) orally with 240 ml of water after an overnight fast, n=6, and matching placebo (2 capsules) orally with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- SAD 6 (Experimental): 600 mg of DM1157 (4 capsules of 150 mg) orally with 240 ml of water after an overnight fast, n=6, and matching placebo (4 capsules) orally with 240 ml of water after an overnight fast, n=2
  Interventions: Drug: DM1157; Other: Placebo
- SAD 7 (Experimental): 900 mg of DM1157 (6 capsules of 150 mg) orally with 240 ml of water after an overnight fast, n=6, and matching placebo (6 capsules) orally with 240 ml of water after an overnight fast (n=2)
  Interventions: Drug: DM1157; Other: Placebo

INTERVENTIONS:
Drug: DM1157 — DM1157 is a novel anti-malarial drug that is derived from chloroquine. DM1157 maintains the efficacy of chloroquine and has molecular features that overcome resistance to chloroquine.
Other: Placebo — Placebo

SUMMARY:
This is a phase 1 trial to evaluate the safety and pharmacokinetics of single and multiple ascending doses and effect of food on the pharmacokinetics of a novel antimalarial drug in healthy adults. The study will enroll 104 healthy volunteers, males and females, aged 18 to 45 years and will consists of 3 parts: Part 1, Single Ascending Dose (SAD); Part 2, Multiple Ascending Dose (MAD); and Part 3, Food Effect. Part 2 and Part 3 may be initiated after a Safety Monitoring Committee (SMC) review and approval of the of Part 1 safety data. Study duration will be 16 months with patient participation duration 14 days for SAD and Food Effect, and 18 days for MAD. The primary objectives of this study are to: 1) assess the safety and tolerability of single doses of DM1157 at levels ranging from 9 mg to 900 mg; 2) assess the safety and tolerability of DM1157 administered as single daily doses for 3 days at levels ranging from 150 mg to 900 mg; 3) assess the safety and tolerability of DM1157 administered with or without food.

DETAILED DESCRIPTION:
This is a first-in-humans, phase 1, randomized, double-blind, single-site, placebo-controlled study in 104 healthy volunteers, males and females, aged 18 to 45 years inclusive. The study will consists of 3 parts: Part 1, Single Ascending Dose (SAD) - participants will be administered a single dose (ranges from 9 mg to 900 mg) of DM1157 orally after fasting or a matching placebo; Part 2, Multiple Ascending Dose (MAD) - participants will be administered three doses (ranges from 150 mg to 900 mg) of DM1157 orally once daily for three days after fasting or a matching placebo; and Part 3, Food Effect - participants will be administered 300 mg of DM1157 orally with high fat meal or a matching placebo. Part 2 and Part 3 may be initiated after a Safety Monitoring Committee (SMC) review and approval of the of Part 1 safety data. Study duration will be 16 months with patient participation duration 14 days for SAD and Food Effect, and 18 days for MAD. The primary objectives of this study are to: 1) assess the safety and tolerability of single doses of DM1157 at levels ranging from 9 mg to 900 mg; 2) assess the safety and tolerability of DM1157 administered as single daily doses for 3 days at levels ranging from 150 mg to 900 mg; 3) assess the safety and tolerability of DM1157 administered with or without food. The secondary objectives are to: 1) assess the PK of single doses of DM1157 at levels ranging from 9 mg to 900 mg, including dose proportionality; 2) assess the PK of DM1157 administered as single daily doses for 3 days at levels ranging from 150 mg to 900 mg; 3) assess the PK of 300 mg DM1157 administered with or without food, including determination of the presence or absence of a food effect on exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or nonpregnant female age 18 to 45 years, inclusive.
2. Can understand the informed consent process and procedures.
3. Agrees to be available for all study visits.
4. If a woman of childbearing potential, agrees to use 2 acceptable contraception methods from 30 days before first study drug administration until 90 days after last study drug administration.

   -Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, or successful Essure(R) placement (permanent, nonsurgical, nonhormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or less than 1 year of the last menses if menopausal.

   -- Includes, but is not limited to, nonmale sexual relationships, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more before the subject receives the first study drug dose, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, or oral contraceptives. If sexually active, methods can include condoms, spermicidal gel, diaphragm, hormonal or nonhormonal intrauterine device, surgical sterilization, oral contraceptive pill, and depot progesterone injections.
5. If male, agrees to use a barrier method of birth control from 30 days before first study drug administration until 90 days after last study drug administration.
6. Has adequate venous access for blood draws.
7. Body mass index (BMI) 18 to 35 kg/m^2, inclusive.

Exclusion Criteria:

1. Any medical disease or condition that, in the opinion of the site PI or appropriate sub investigator, is a contraindication to study participation.
2. History of clinically significant ECG abnormalities or has clinically significant ECG abnormalities at Screening.
3. Use of any prescription medication (excluding oral contraceptive pills in females) within 14 days before first study drug administration.
4. Use of occasional nonprescription drugs (oral or topical) within 7 days before first study drug administration unless permitted by the investigator.

   - Nonprescription drugs include vitamins, antacids, herbal or dietary supplements, and topical gels, creams, etc., that in the opinion of the site PI could interfere with the study drug.
5. Hypertension with confirmed systolic blood pressure (BP) greater than 145 mm Hg or confirmed diastolic BP greater than 90 mm Hg, measured after 10 to 15 minutes of rest.
6. Heart rate (HR) less than 50 bpm or greater than 100 bpm.
7. Body weight less than 50 kg.
8. History of a significant illness within 2 weeks before dosing (subjects can screen after illness is resolved for 2 weeks).
9. History of hemolytic anemia.
10. History of retinal eye disease.
11. History of hearing loss.
12. History of seizures.
13. History of thyroid disease or currently on replacement therapy for hypothyroidism.
14. History of liver disease other than Gilbert's syndrome.
15. History of severe drug hypersensitivity, including a severe allergic reaction, anaphylaxis, or convulsions following any medication, vaccination, or infusion.
16. History of malignancy except low-grade skin cancer (ex. basal cell carcinoma thought to be cured).
17. Known diagnosis of prolonged QT interval, congenital long QT syndrome, bradyarrhythmias, or uncompensated heart failure.
18. History of drug or alcohol abuse within 12 months before Screening.
19. History of renal disease.
20. Excessive consumption of beverages containing xanthine bases, including Red Bull, chocolate, etc., or more than 400 mg of caffeine per day (more than 4 cups of coffee per day).
21. Consumption of citrus fruits or juices (ex. pomegranate, orange, lime, grapefruit) within 7 days before first study drug administration.
22. Use of nicotine-containing products within 30 days before Screening and until completion of study.
23. Consumption of alcohol within 24 hours of first study drug administration.
24. Has any condition or disease that might affect drug absorption, distribution, or excretion (ex. gastrectomy, diarrhea).
25. Positive serology results for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody.
26. Positive drug screen (cannabinoids, amphetamines, barbiturates, cocaine, opiates, benzodiazepines, phencyclidine) or positive breathalyzer test for alcohol.

    - Subjects should be notified by phone not to consume any poppy seeds within 24 hours before the Screening blood test to avoid false a positive opioid test result.
27. History of allergic reaction or intolerance to CQ.
28. Males with a QTcF greater than 450 ms or females with a QTcF greater than 460 ms (Fridericia's correction) at Screening.
29. Positive pregnancy test within 24 hours before study drug administration; pregnant or nursing.
30. Screening lab tests, specifically total WBC, platelet count, hemoglobin, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and creatinine, which meet Grade 1 or higher toxicity. Safety laboratory tests drawn on Day -1 will serve as baseline. Day -1 safety laboratory tests with a Grade 1 severity will not exclude a subject from participation if assessed as not clinically significant by the PI or designee.
31. Any specific condition that, in the judgment of the site PI, precludes participation because it could affect subject safety.
32. Received an experimental agent within 30 days or 5 half-lives (whichever is longer) before study drug administration.

    - Vaccine, drug, biologic, device, blood product, or medication
33. Is participating or plans to participate in another clinical study with an interventional agent that will be received during participation in this study.
34. Has donated more than 500 mL of blood within the last month before Screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Count of participants who discontinued single ascending dose (SAD) for safety reasons | Day 1 through Day 14
Occurrence of abnormal ECG changes from baseline (categorized as clinical Adverse Events (AEs)) for a single dose taken after food ingestion | Day 1 through Day 14
Occurrence of abnormal ECG changes from baseline (categorized as clinical Adverse Events (AEs)) for multiple ascending dose (MAD) | Day 1 through Day 18
Occurrence of abnormal ECG changes from baseline (categorized as clinical Adverse Events (AEs)) for single ascending dose (SAD) | Day 1 through Day 14
Occurrence of abnormal vital sign changes from baseline (categorized as clinical Adverse Events (AEs)) for a single dose taken after food ingestion | Day 1 through Day 14
Occurrence of abnormal vital sign changes from baseline (categorized as clinical Adverse Events (AEs)) for multiple ascending dose (MAD) | Day 1 through Day 18
Occurrence of abnormal vital sign changes from baseline (categorized as clinical Adverse Events (AEs)) for single ascending dose (SAD) | Day 1 through Day 14
Occurrence of Adverse Events (AE) for a single dose taken after food ingestion | Day 1 through Day 14
Occurrence of Adverse Events (AE) for multiple ascending dose (MAD) | Day 1 through Day 18
Occurrence of Adverse Events (AE) for single ascending dose (SAD) | Day 1 through Day 14
Occurrence of laboratory Adverse Events (AE) for a single dose taken after food ingestion | Day 1 through Day 14
Occurrence of laboratory Adverse Events (AE) for multiple ascending dose (MAD) | Day 1 through Day 18
Occurrence of laboratory Adverse Events (AE) for single ascending dose (SAD) | Day 1 through Day 14

SECONDARY OUTCOMES:
Plasma levels of a single dose of DM1157 taken after food ingestion | Day 1 through Day 14
Plasma levels of multiple ascending dose (MAD) of DM1157 | Day 1 through Day 18
Plasma levels of single ascending dose (SAD) of DM1157 | Day 1 through Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Medicine - Duke Clinical Research Institute - Duke Clinical Research Unit, Durham, North Carolina, United States

REFERENCES:
- [Derived] Balevic SJ, Raja SM, Randell R, Deye GA, Conrad T, Nakamura A, Peyton DH, Shotwell S, Liebman K, Cohen-Wolkowiez M, Guptill JT. Adverse Reactions in a Phase 1 Trial of the Anti-Malarial DM1157: An Example of Pharmacokinetic Modeling and Simulation Guiding Clinical Trial Decisions. Infect Dis Ther. 2022 Apr;11(2):841-852. doi: 10.1007/s40121-022-00605-z. Epub 2022 Feb 20. PMID 35184256